CLINICAL TRIAL: NCT03229343
Title: Impact of a Systematic Palliative Care on Quality of Life, in Advanced Idiopathic Pulmonary Fibrosis (IPF). A Randomized Multi-center Trial.
Brief Title: Impact of a Systematic Palliative Care on Quality of Life, in Advanced Idiopathic Pulmonary Fibrosis.
Acronym: PALIF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P150965
Record Dates: First submitted 2017-07-04; First posted 2017-07-25 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2017-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: idiopathic pulmonary fibrosis, palliative care
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Experimental arm : supportive care, systematic and joint to pneumological consultation, monthly, starting at M0 and continuing up to M6.
  Non interventionnel arm: only pneumological consultation performed at M0, M3 and M6.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Supportive care, systematic and joint to pneumological consultation, monthly, starting at M0 and continuing up to M6.
  Interventions: Other: Supportive care
- standard (No Intervention): pneumological consultation performed at M0, M3 and M6

INTERVENTIONS:
Other: Supportive care — supportive care, systematic and joint to pneumological consultation, monthly, starting at M0 and continuing up to M6.
  Arms: Experimental

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a rare and severe disease with a survival median between 2 and 4 years which leads to a profound alteration of the quality of life.

In thoracic oncology, the systematic and early intervention of a palliative care team result in an improvement of quality of life for patients.

In the princeps study published in 2010, the early intervention of a dedicated palliative care team was compared to standard care in a randomized trial of 150 patients and shows a significant improvement : (i) of quality of life (main objective), (ii) of depression scores and even overall survival (11.6 months vs. 8.9 months, P = 0.02), (iii) a benefit in terms of understanding the diagnosis and therapeutic goals (3), (iv) diminution of adapted hospitalization in end of life (in emergency or not).

Considering some analogy points between IPF and advanced lung cancer (prognosis, respiratory symptom, psychological burden), it seemed reasonable to assume that the joint systematic intervention of chest physician and palliative care team may provide a significant benefit in terms of quality of life for patients with severe IPF.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a rare and severe disease with a survival median between 2 and 4 years which leads to a profound alteration of the quality of life. This alteration results from different consequences of the IPF: progressive shortness of breath, irritative cough refractory to treatments, exhaustion, limitation of activity, social isolation, and psychic consequences such as fear, anxiety and depression.

The only current curative treatment of the disease is pulmonary transplantation, but it's only feasible for a minority of patients. Anti-fibrotic drugs, such as pirfenidone and nintedanib, are likely to slow the progression of IPF but have no impact on patients' quality of life.

The symptomatic treatment aimed at relieving respiratory discomfort and the patient's quality of life is therefore fundamental, and the IPF meets in many ways the challenges of lung cancer.

In thoracic oncology, the systematic and early intervention of a palliative care team result in an improvement of quality of life for patients.

In the princeps study published in 2010, the early intervention of a dedicated palliative care team was compared to standard care in a randomized trial of 150 patients and shows a significant improvement : (i) of quality of life (main objective), (ii) of depression scores and even overall survival (11.6 months vs. 8.9 months, P = 0.02), (iii) a benefit in terms of understanding the diagnosis and therapeutic goals (3), (iv) diminution of adapted hospitalization in end of life (in emergency or not).

Considering some analogy points between IPF and advanced lung cancer (prognosis, respiratory symptom, psychological burden), it seemed reasonable to assume that the joint systematic intervention of chest physician and palliative care team may provide a significant benefit in terms of quality of life for patients with severe IPF.

Objective:

To investigate the benefit on quality of life, evaluated after 6 months, of a systematic, formalized and joint intervention of a palliative intervention staff and a chest physician team compared to standard care for patients with severe IPF.

Secondary endpoints

1. To evaluate the benefit of the systematic, formalized and joint intervention of a palliative care team and a chest physician team on:

   * Mood and depression
   * Understanding of diagnosis and therapeutic objectives, frequency of drafting of advance directives regarding end-of-life
   * Respiratory symptoms (cough and dyspnea)
   * The course of care, the use of palliative care stays and the duration of hospital stays (number and duration of hospitalizations).
   * Overall survival and place of death.
2. Carry out a medico-economic study evaluating the incremental cost-utility and cost-effectiveness ratio (overall survival criterion)

ELIGIBILITY:
Inclusion Criteria:

* Age> 40 years
* Patient with confirmed diagnosis of IPF according to the American Thoracic Society (ATS) / European Respiratory Society (ERS) / Japanese Respiratory Society (JRS) / Latin American Thoracic Association (ALAT) criteria. The patient may be included regardless of the date of diagnosis.
* Advanced IPF with Forced Vital Capacity (FVC) <50%" of predicted value and / or Diffusing capacity for carbon monoxide ((DLCO) <30% of predicted value or inability to achieve the Functional Respiratory Investigations (EFR) due to respiratory severity. EFR dated less than 3 months.
* Absence of argument for acute or subacute exacerbation in the last 6 months.
* Patient who can be followed in ambulatory consultation/ outpatient consultation.
* Informed consent signed (signed by the patient or in the presence of a third party for patients who are poorly fluent in French).
* Affiliation to the social security system.

Exclusion Criteria:

* Patient unable to respond to quality of life questionnaires.
* Inability (physical or mental) to give a written informed consent.
* Acute exacerbation of fibrosis in the previous 6 months.
* Patient eligible for a pulmonary transplant.
* Participation in other therapeutic trial
* Patient cannot be followed in ambulatory consultation.
* Patient under trustee

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
The benefit of a systematic, formalized and joint intervention of a palliative intervention staff and a chest physician team on quality of life, evaluated after 6 months by the Short Form (36) Health Survey. | at 6 months after inclusion
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The Short Form (36) Health Survey consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health. This score has already been used for IPF

SECONDARY OUTCOMES:
The benefit of the systematic, formalized and joint intervention of a supportive care and a pneumologist team on the benefit of the systematic, formalized and joint intervention of a supportive care and a pneumologist team on Mood and depression | at 3 and 6 months after inclusion
  evaluated by the Hospital Anxiety and Depression questionnaire.
  * Understanding of diagnosis and therapeutic objectives, frequency of drafting of advance directives
  * Respiratory symptoms (dyspnea)
  * The course of care, the use of palliative care stays and the duration of hospital stays (number and duration of hospitalizations).
  * Overall survival and place of death.
The benefit of the systematic, formalized and joint intervention of a supportive care and a pneumologist team on Understanding of diagnosis and therapeutic objectives, frequency of drafting of advance directives. | at 3 and 6 months after inclusion
  the benefit of the systematic, formalized and joint intervention of a supportive care and a pneumologist team on Understanding of diagnosis and therapeutic objectives, frequency of drafting of advance directives will be evaluated by the illness understanding questionnaire.
The benefit of the systematic, formalized and joint intervention of a supportive care and a pneumologist team on Respiratory symptoms (dyspnea) | at 3 and 6 months after inclusion
  The benefit of the systematic, formalized and joint intervention of a supportive care and a pneumologist team on Respiratory symptoms (dyspnea) will be evaluated by St George's respiratory questionnaire (SGRQ) and Transition Dyspnea Index (TDI)
The benefit of the systematic, formalized and joint intervention of a supportive care and a pneumologist team on the course of care. | at 3 and 6 months after inclusion
  the benefit of the systematic, formalized and joint intervention of a supportive care and a pneumologist team on the course of care, the use of palliative care stays and the duration of hospital stays (number and duration of hospitalizations)
The benefit of the systematic, formalized and joint intervention of a supportive care and a pneumologist team on the Overall survival. | between inclusion and date of death or last news. (survival follow-up visit at month 12)
  the benefit of the systematic, formalized and joint intervention of a supportive care and a pneumologist team on the Overall survival measured between inclusion and date of death or last news.
Carry out a medico-economic study evaluating the incremental cost-utility and cost-effectiveness ratio (overall survival criterion) | at 3 and 6 months after inclusion
  This outcome is evaluated by the medico-economic questionnaire : EuroQol five dimensions questionnaire (EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Duchemann, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (11):
- France (11):
  - Centre Hospitalier Robert Ballanger, Aulnay-sous-Bois
  - Hôpital Avicenne, Bobigny
  - Centre Hospitalier de Versailles Andre Mignot, Le Chesnay
  - Hôpital LOUIS PRADEL, Lyon
  - Hôpital NORD, Marseille
  - Hôpital MARC JACQUET, Melun
  - Hôpital GEORGES POMPIDOU (HEGP), Paris
  - Hôpital Tenon, Paris
  - Hôpital Pontchaillou, Rennes
  - Hôpital DELAFONTAINE, Saint-Denis
  - Hôpital LARREY, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swigris JJ, Brown KK, Behr J, du Bois RM, King TE, Raghu G, Wamboldt FS. The SF-36 and SGRQ: validity and first look at minimum important differences in IPF. Respir Med. 2010 Feb;104(2):296-304. doi: 10.1016/j.rmed.2009.09.006. Epub 2009 Oct 7. PMID 19815403
- [Background] Swigris JJ, Kuschner WG, Jacobs SS, Wilson SR, Gould MK. Health-related quality of life in patients with idiopathic pulmonary fibrosis: a systematic review. Thorax. 2005 Jul;60(7):588-94. doi: 10.1136/thx.2004.035220. PMID 15994268
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875